CLINICAL TRIAL: NCT04315415
Title: A Histological Study Evaluating Silk Voice and Crosslinked Hyaluronic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofregen Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SOF-003
Record Dates: First submitted 2020-02-20; First posted 2020-03-19 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Vocal Fold Palsy; Vocal Cord Paralysis; Vocal Cord Atrophy
Keywords: silk, vocal fold
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Intervention Model Description: Each subject enrolled will receive implantation of both Silk Voice and control material.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 6 month explant (Other): Silk Voice and control material are implanted. The implanted material is explanted at 6 months.
  Interventions: Device: Silk Voice
- 12 month explant (Other): Silk Voice and control material are implanted. The implanted material is explanted at 12 months.
  Interventions: Device: Silk Voice
- 24 month explant (Other): Silk Voice and control material are implanted. The implanted material is explanted at 24 months.
  Interventions: Device: Silk Voice

INTERVENTIONS:
Device: Silk Voice — Silk Voice comprised of silk protein and cross-linked hyaluronic acid (HA)

SUMMARY:
The primary study goal is to evaluate the histological characteristic of Silk Voice to evaluate the potential for Silk Voice to deliver long-term results to patients.

DETAILED DESCRIPTION:
The primary study goal is to evaluate the histological characteristic of Silk Voice at a surrogate implantation site to evaluate the potential for Silk Voice to deliver long-term results to patients. Information obtained from this study will help clinician determine Silk Voice's treatment duration and whether Silk Voice is appropriate for their patient.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for enrollment, the Subject must meet the following:

  * males or non-pregnant, non-breastfeeding females 21 to 65 years old who are willing to comply with the requirements of the study, including sequential photography, periodic check-ins and retrieval of implanted materials;
  * women of childbearing potential using an acceptable form of birth control during the study period and willingness to take a urine pregnancy test at baseline and at the biopsy date;
  * sign the Informed Consent form and the Authorization for Use and Release HIPAA form prior to any study-related procedures being performed.
  * read and understand English

Exclusion Criteria:

* Patients will not enroll in the study if they meet any of the following exclusion criteria:

  * a history of allergy or hypersensitivity to injectable hyaluronic acid gel;
  * a history of allergy or hypersensitivity to silk;
  * a history of severe allergies manifested by a history of anaphylaxis or history or presence of multiple severe allergies
  * history of allergies of lidocaine
  * a history of susceptibility to keloid formation, hypertrophic scarring, and pigmentation disorders.
  * currently have a hyaluronic acid device implanted
  * the presence of any contraindication to the implant procedures, including use of platelet inhibiting agents or other anticoagulant, in a relevant period before study entry (per the treating investigator's judgment);
  * the presence of any condition, which in the opinion of the investigator, that makes the subject unable to complete the study per protocol;
  * the presence of known allergies or hypersensitivity reactions to local topical anesthetics or nerve blocking agents (if such products are intended to be used for that subject);
  * the presence of cancerous or pre-cancerous lesions in the area to be treated;
  * the presence of moderate or severe abnormal rating for firmness or detection of any abnormal structure at the site of injection, such as a scar or lump;
  * the current use of immunosuppressive therapy;
  * who are using substances that can prolong bleeding (such as aspirin, nonsteroidal anti-inflammatory drugs, and warfarin) may, as with any injection, experience increased bruising or bleeding at treatment sites
  * a history of connective tissue diseases such as rheumatoid arthritis, systemic lupus erythematosus, polymyositis, dermatomyositis or scleroderma;
  * participation in any interventional clinical research study within 30 days prior to randomization;
  * subjects not likely to stay in the study for up to 13 months because of other commitments, concomitant conditions, or past history;
  * subjects anticipated to be unreliable; or subjects who have a concomitant condition that might confuse or confound study treatments or assessments;
  * Subject with skin conditions (discoloration, textured, scarring, etc.) in postauricular region that may complicate study evaluation metrics
  * Subjects that are not considered to be an appropriate candidate at the discretion of the investigator.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Number of subjects exhibiting histological evidence of newly deposited tissue compared to control implantation. | 6 month
  Tissue samples extracted at 6 -month time points will be qualitatively evaluated for presence of tissue deposition. Changes in tissue composition will be assessed.
Number of subjects exhibiting histological evidence of newly deposited tissue compared to control implantation. | 12 month
  Tissue samples extracted at 12 -month time points will be qualitatively evaluated for presence of tissue deposition. Changes in tissue composition will be assessed.
Number of subjects exhibiting histological evidence of newly deposited tissue compared to control implantation. | 24 month
  Tissue samples extracted at 24 -month time points will be qualitatively evaluated for presence of tissue deposition. Changes in tissue composition will be assessed.

SECONDARY OUTCOMES:
Number of patient and number of reported adverse events reported | 6 month
  Localized adverse event associated with material implantation. The number of patients and type of adverse events will be evaluated.
Number of patient and number of reported adverse events reported | 12 month
  Localized adverse event associated with material implantation. The number of patients and type of adverse events will be evaluated.
Number of patient and number of reported adverse events reported | 24 month
  Localized adverse event associated with material implantation. The number of patients and type of adverse events will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- DeNova Research, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No